CLINICAL TRIAL: NCT00729365
Title: Nocturnal Hypertension and Prevention of Microalbuminuria in Type 1 Diabetes
Brief Title: PREVENTKD (Prevent Risks by Early interVEntion at Nighttime in Type 1 Diabetes for Kidney Disease)
Acronym: PREVENTKD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data from other studies showed that study could not be completef successfully
Sponsor: Northwestern University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mark Molitch, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1U01DK071733-01A1 (NIH); 1U01DK071733-01A1 (NIH)
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes
Keywords: Urine albumin excretion rates; Nighttime and daytime blood pressure; Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dippers - Placebo Treated (Placebo Comparator): Subjects with normal nighttime blood pressure profile that decreases at night (Dippers). This group are all given placebo.
  Interventions: Drug: Placebo
- NonDippers - Placebo Treated (Placebo Comparator): Subjects with nighttime blood pressure that does not drop during the night (non-dippers). This group will be given placebo.
  Interventions: Drug: Placebo
- NonDippers - Ramipril Treated (Active Comparator): Subjects with nighttime blood pressure that does not drop during the night (non-dippers). This group will be given ACE inhibitor (study medication).
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — ACE inhibitor known as Ramipril
  Subjects with nighttime blood pressure that does not drop during the night ("non-dippers") maybe randomized into this group and given an ACE inhibitor (study medication). Therefore, the "Non-Dippers" groups II and III will be randomized to receive either drug or placebo.
  Other Names: ACE Inhibitor
  Arms: NonDippers - Ramipril Treated
Drug: Placebo — Dippers (category of subjects with a nighttime dip in blood pressure) will all be given Placebo. Control group.
  Arms: Dippers - Placebo Treated
Drug: Placebo — Subjects with nighttime blood pressure that does not drop during the night ("non-dippers") maybe randomized into the control group and given Placebo.
  Arms: NonDippers - Placebo Treated

SUMMARY:
The purpose of this study is to determine if the early treatment with a blood pressure medication (an ACE Inhibitor) can prevent or delay the development of kidney disease (microalbuminuria) in patients with Type 1 diabetes who have normal blood pressure and urine albumin levels.

DETAILED DESCRIPTION:
Only a fraction of persons with Type 1 diabetes (less than 40%) develop diabetic kidney disease (nephropathy). When the urinary albumin (a protein normally excreted in small amounts) is within the normal range, the prevalence of high blood pressure (hypertension) based on office blood pressure readings is very low. Many of these persons, however, develop nocturnal hypertension (high nighttime blood pressure) before the development of abnormally high urinary albumin excretion (a condition referred to as microalbuminuria). Currently, early treatment with medications called ACE inhibitors is only recommended after there is an indication of kidney damage, as reflected by the presence of microalbuminuria. Beginning ACE inhibitor therapy is currently not recommended prior to the development of microalbuminuria, unless patients have high blood pressure, because it would result in over-treatment of many people. By the time that microalbuminuria develops, however, kidney damage may be present and many patients will develop kidney disease. It would therefore be beneficial to identify those subjects who will develop microalbuminuria, so that treatment could be started early for those individuals. Persons who may go on to develop protein in their urine and eventual kidney disease perhaps could be identified on the basis of an abnormal fall (too little) in blood pressure at night. This pattern should not be confused with high blood pressure, but instead seen as an early indication present before the development of high blood pressure and microalbuminuria.

The purpose of the current study is therefore aimed at demonstrating that it is possible to prevent kidney disease in patients with type 1 diabetes and normal office blood pressure and urine protein excretion by selecting them on the basis of an abnormal fall in blood pressure at night. Moreover, this clinical trial will reveal the impact of long-term administration of an ACE inhibitor on nighttime blood pressure and also assess changes in the relative stiffness of blood vessels(endothelial dysfunction) in persons with type 1 diabetes over time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 diabetes confirmed by C peptide measurements.
* Male and Female subjects of all races will be included in this study.
* Subjects age must be between 13 to 50 years
* Duration of the disease (from time of diagnosis of diabetes) must be between 5 to 28 years.
* Subjects must be normotensive defined as a systolic blood pressure of ≤ 130 mmHg and diastolic of ≤ 85 mmHg in subjects 18 and older and for children (ages 13-17) blood pressure will be in the normal range based on standard tables which takes in to account gender, height and age.
* The mean 24 blood pressure must meet the same criteria as the office blood pressures outlined above.
* Subject must have normoalbuminuria (UAE < 30 mg/24 hrs)
* If subject is a female she must not be breast-feeding, and not of child-bearing potential, defined as post-menopausal for at least 1 year or surgically sterile; if she is of child bearing potential, then she must be practicing one of the following methods of birth control: 1) condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD), 2) contraceptives (oral or parenteral) initiated three months prior to study drug administration, 3) maintain a monogamous relationship with a vasectomized partner, or 4) total abstinence from sexual intercourse.

Exclusion Criteria:

* Type 2 diabetics and other types of diabetics such as those with maturity onset diabetes or the young (MODY) will be excluded on the basis of established clinical criteria.
* Subjects who have a history of hypertension or is taking any hypertensive medications.
* Females who are pregnant or express a desire to become pregnant during the study. Females who are breast-feeding. Refer to details in inclusion criteria above regarding females.
* Subjects who have a history of taking ACE inhibitors within the last six months or have a current indication for ACE inhibitor therapy.
* Subjects (18 years of age and over) with a current blood pressure above 130mmHg/85mmHg. Subjects (13-17 years of age) who do not meet the normal range based on the standard tables
* Subjects who are currently microalbuminuric i.e. 24hr albumin > 30mg
* Subjects who have participated in an interventional clinical trial involving ABPM 6 months prior to this study.
* Subjects that have a diagnosis of chronic atrial fibrillation.
* Subjects with a lifestyle that would disrupt normal circadian rhythm (i.e. night-shift workers).
* Subjects with a current serious co-morbid condition for which life expectancy is <2 years.
* Subjects with a history of non-compliance, or psychiatric disturbance that would preclude successful completion of the study.
* Inability to give informed consent.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Molitch, MD, Principal Investigator — Professor of Medicine
Locations (6):
- United States (6):
  - University of Florida, Gainesville, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Endocrinology Section, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois

REFERENCES:
- [Background] Lurbe E, Redon J, Kesani A, Pascual JM, Tacons J, Alvarez V, Batlle D. Increase in nocturnal blood pressure and progression to microalbuminuria in type 1 diabetes. N Engl J Med. 2002 Sep 12;347(11):797-805. doi: 10.1056/NEJMoa013410. PMID 12226150
- [Background] Dolan E, Stanton A, Thijs L, Hinedi K, Atkins N, McClory S, Den Hond E, McCormack P, Staessen JA, O'Brien E. Superiority of ambulatory over clinic blood pressure measurement in predicting mortality: the Dublin outcome study. Hypertension. 2005 Jul;46(1):156-61. doi: 10.1161/01.HYP.0000170138.56903.7a. Epub 2005 Jun 6. PMID 15939805
- [Background] Lurbe A, Redon J, Pascual JM, Tacons J, Alvarez V, Batlle DC. Altered blood pressure during sleep in normotensive subjects with type I diabetes. Hypertension. 1993 Feb;21(2):227-35. doi: 10.1161/01.hyp.21.2.227. PMID 8428785
- [Background] Haller MJ, Stein J, Shuster J, Theriaque D, Silverstein J, Schatz DA, Earing MG, Lerman A, Mahmud FH. Peripheral artery tonometry demonstrates altered endothelial function in children with type 1 diabetes. Pediatr Diabetes. 2007 Aug;8(4):193-8. doi: 10.1111/j.1399-5448.2007.00246.x. PMID 17659060

RESULTS

PARTICIPANT FLOW:
Groups:
- Dippers - Placebo Group: Subjects with normal nighttime blood pressure profile that decreases at night (Dippers). This group are all given placebo.
  Placebo: Dippers (category of subjects with a nighttime dip in blood pressure) will all be given Placebo. Control group.
- Non-dippers - Placebo: Subjects with nighttime blood pressure that does not drop during the night (non-dippers). This group will be given placebo.
  Placebo: Subjects with nighttime blood pressure that does not drop during the night ("non-dippers") maybe randomized into the control group and given Placebo.
- Non-Dippers - Ramipril: Subjects with nighttime blood pressure that does not drop during the night (non-dippers). This group will be given ACE inhibitor (study medication).
  Ramipril: ACE inhibitor known as Ramipril
  Subjects with nighttime blood pressure that does not drop during the night ("non-dippers") maybe randomized into this group and given an ACE inhibitor (study medication). Therefore, the "Non-Dippers" groups II and III will be randomized to receive either drug or placebo.
Period: Overall Study
Arm/Group | Dippers - Placebo Group | Non-dippers - Placebo | Non-Dippers - Ramipril
Started | 33 | 6 | 7
Completed | 0 (Study terminated) | 0 (Study Terminated) | 0 (Study terminated)
Not Completed | 33 | 6 | 7
Not completed — Physician Decision | 33 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Dippers - Placebo: Subjects with normal nighttime blood pressure profile that decreases at night (Dippers). This group are all given placebo.
  Placebo: Dippers (category of subjects with a nighttime dip in blood pressure) will all be given Placebo. Control group.
- Total: Total of all reporting groups
Arm/Group | Dippers - Placebo | Non-Dippers - Placebo | Non-Dippers - Ramipril | Total
Number analyzed (Participants) | 33 | 6 | 7 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 2
  Between 18 and 65 years | 32 | 5 | 7 | 44
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 30.0 [13 to 49] | 27.5 [17 to 44] | 30.0 [23 to 47] | 29.5 [13 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 6 | 4 | 32
  Male | 11 | 0 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 6 | 7 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 28 | 5 | 7 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 33 | 6 | 7 | 46

OUTCOME MEASURES:

1. Primary Outcome: Development of Microalbuminuria (High Urine Albumin). Hypertension, Urine and Blood Markers Will Also be Evaluated for Assessment of Kidney Disease State.
Time Frame: at 3months and then every 6months during the 5years of the study
Arm/Group | Dippers - Placebo Group | Non-dippers - Placebo | Non-Dippers - Ramipril
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: We Will Assess Changes in the Relative Stiffness of Your Arteries (Endothelial Dysfunction) in Persons With Type 1 Diabetes Over the 5year Study.
Time Frame: year 1, 3, 5 and after the washout phase (5years and 1month)
Arm/Group | Dippers - Placebo | Non-Dippers - Placebo | Non-Dippers - Ramipril
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dippers - Placebo | Non-Dippers - Placebo | Non-Dippers - Ramipril
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely because of new information from the literature from other studies showing that this study could not be successful.

Only 59 patients were screened and consented and 46 were found acceptable who were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No